CLINICAL TRIAL: NCT04740684
Title: Microbiome Individuality and Stability Over Time
Acronym: MISO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Timothy Meyer, Professor of Nephrology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 44718
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Diet

STUDY DESIGN:
Intervention Model Description: All participants will consume the exact same diet for one week. Samples will be collected before, during and after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standardized diet — Standardized diet is prepared in a commercial kitchen and packaged in single serve portions to provide to participants to consume for 7 days

SUMMARY:
Microbial derived uremic solutes (p-cresol sulfate, indoxyl sulfate, and phenylacetylglutamine) are present in blood and excreted into the urine. Uremic solutes have high inter-individual variability of unclear etiology, that the investigators hypothesize is due to intestinal microbiome variation and/or dietary variation between people. In this study, the investigators will collect baseline samples on participant's habitual diet. The investigators will then administer a homogenous diet to all participants for 7 days and examine levels of uremic solutes in the urine via 24-hour urine collection during this period. In parallel, the investigators will monitor microbiome composition. The investigators predict that during the period subjects are consuming the same, homogenous diet, their excretion of uremic solutes (p-cresol sulfate, indoxyl sulfate, and phenylacetylglutamine) into the urine will have less inter-individual variation.

DETAILED DESCRIPTION:
Participants will be asked to eat exactly the same meal for one week and to eat this same meal three times each day. Subjects will be allowed to eat as much of this meal as they want and to eat enough so that they do not lose weight. The food will provide a nutritionally adequate diet, designed by a registered dietitian. Participants will be asked not to eat anything else including candy, snacks, etc. and not to drink anything except water including coffee, tea, sodas, or alcoholic drinks.

Samples will be collected at 5 time points:

2 weeks prior to starting test diet, Baseline (day 1 on diet), day 4 on the diet, day 7 on the diet, 7 days after end of diet.

Samples collected include:

Blood sample Stool sample 24 hr urine collection Diet and Gastrointestinal questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

Exclusion Criteria:

* pregnancy
* diabetes
* gastrointestinal disease
* use of medications thought by the investigators to have a significant effect on the microbiome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Uremic solute variability | 2 years
  25% reduction of the coefficient of variation of 24hr urinary excretion of at least 1 of 3 uremic solutes (p-cresol sulfate, indoxyl sulfate or phenylacetylglutamine) measured in mg/day/1.73 during the homogenous diet period as compared to the baseline/habitual diet period.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States